CLINICAL TRIAL: NCT03838328
Title: Dose Effect of Tranexamic Acid on the Incidence of Deep Venous Thrombus in Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Dose Effect of Tranexamic Acid on the Incidence of Deep Venous Thrombus in Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SHI Jia (Other)
Responsible Party: Sponsor-Investigator, SHI Jia, Associate Professor and Vice Chair of the Anesthesiology Department, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dose effect of TA on DVT
Record Dates: First submitted 2019-02-01; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Thromboses, Deep Vein; Tranexamic Acid Adverse Reaction
Keywords: dose effect; tranexamic acid; deep vein thromboses
MeSH Terms: conditions — Venous Thrombosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation is masked for the participant, care provider, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose group 1 (Experimental): The dose regimen of tranexamic acid in group 1 includes a loading dose of 30mg/kg before skin incision and a maintenance dose of 20mg/kg/hr until the end of the operation.
  Interventions: Drug: Tranexamic Acid
- Dose group 2 (Experimental): The dose regimen of tranexamic acid in group 2 includes a loading dose of 20mg/kg before skin incision and a maintenance dose of 15mg/kg/hr until the end of the operation.
  Interventions: Drug: Tranexamic Acid
- Dose group 3 (Active Comparator): The dose regimen of tranexamic acid in group 3 includes a loading dose of 10mg/kg before skin incision and a maintenance dose of 10mg/kg/hr until the end of the operation.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid will be delivered by loading dose plus maintenance infusion until the end of the operation.

SUMMARY:
In recent years, the lysine analogs tranexamic acid (TXA) has gained wide use in cardiac surgery as a blood-sparing agent. However, the safety of the drug and its impact on overall outcomes of cardiac surgery remains debated. The current study evaluates the dose effect of TXA on the incidence of deep venous thrombus (DVT) in cardiac surgery with cardiopulmonary bypass. Also, the dose effect of TXA on bleeding and allogeneic transfusion is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving selective cardiac surgery with cardiopulmonary bypass due to coronary, valvular or congenital heart disease
* Written consent obtained

Exclusion Criteria:

* Allergy or contraindication to tranexamic acid
* Severe renal impairment (serum creatinine >250 μmol/l, or estimated creatinine clearance <25 ml/min)
* Thromboembolic disease including but not limited to: history of pulmonary embolism, spontaneous arterial thrombosis or familial hypercoaguability (eg. Lupus anticoagulant, protein C deficiency)
* Thrombocytopenia defined as a platelet count <100,000/ml
* Coagulopathy defined as an international normalized ratio > 1.5 prior to surgery
* Currently enrolled in another perioperative interventional study
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of deep venous thrombosis | Within 7 days postoperatively
  Defined as the incidence of new-onset deep venous thrombosis postoperatively diagnosed by ultrasound

SECONDARY OUTCOMES:
The rate of new-onset thrombotic events | Within 90 days postoperatively
  Thrombotic events include ischemic stroke, renal failure, myocardial infarction and pulmonary embolism
The rate of allogeneic RBC transfusion | Within 30 days postoperatively
  Allogeneic blood product includes packed red blood cell
The volume of allogeneic RBC transfusion | Within 30 days postoperatively
  Allogeneic blood product includes packed red blood cell
Length of stay in ICU and hospital | Within 90 days postoperatively
  The time interval between the end of the operation and the discharge from ICU or the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shi, M.D., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences， Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No